CLINICAL TRIAL: NCT06815458
Title: The Effect of Reflective Learning Based on Visual Mind Mapping on Developing Knowledge and Skills Regarding Vital Signs in Nursing Education: a Randomized Controlled Trial
Brief Title: Visual Mind Mapping in Nursing Education
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 10
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Education
Keywords: Mind Mapping; Nursing students; Vital signs
MeSH Terms: interventions — Nursing Education Research

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Nursing education — Mind mapping based learning

SUMMARY:
Visual Mind Mapping in Nursing Education

DETAILED DESCRIPTION:
In this study, by using both teaching strategies in an integrated manner, it is aimed for students to grasp the information in depth and use this information effectively in a clinical environment instead of just superficial learning. The originality of the study is that it is about vital signs with first-year nursing students. It is anticipated that the study will contribute to the literature in terms of the development of knowledge-based skills such as pulse, respiration, blood pressure and body temperature.

ELIGIBILITY:
Inclusion Criteria:

* Receiving training on vital signs for the first time
* Being a first-year nursing student

Exclusion Criteria:

* Having previously received training on vital signs
* Having class absences, not taking the final and follow-up tests

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nursing students
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The effect of education provided with mind mapping on success in nursing students | 01/11/2024-31/12/2024
  Nursing education

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)